CLINICAL TRIAL: NCT06755957
Title: Investigation of the Effectiveness of Wall Angels Exercise Combined With Standard Exercises in Young Adults With Kyphotic Posture: A Double-Blind Randomized Controlled Trial
Brief Title: Effectiveness of Standard Exercises and Wall Angels Exercise in Young Adults With Kyphotic Posture
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Mesut ERGAN, Assistant Professor, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-27-2024/80/4
Record Dates: First submitted 2024-12-13; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Kyphosis Thoracic; Exercise Therapy
Keywords: Corrective Exercise; Kyphosis; Posture; Thoracic Mobility
MeSH Terms: conditions — Kyphosis | interventions — Exercise; Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): 1. Posture Exercises (3 sets * 15 reps):
  1a) Shoulder lift
  1b) Shoulder forward circles
  1c) Shoulder backward circles 2. Pectoral Stretch Exercise (3 sets * 10 reps; each stretch held for 30 seconds; for right and left sides) 3. Back Strengthening Exercise (3 sets * 15 reps) 4. Self Mobilization Exercise (3 sets * 10 reps; for right and left sides) 5. Cat-Camel Exercise (3 sets * 10 reps) 6. Breathing Exercises (3 sets * 10 reps): 6a) Diaphragmatic breathing 6b) Segmental breathing 7. Wall angels exercise (2 sets * 10 reps)
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION
- Control arm (Active Comparator): 1. Posture Exercises (3 sets * 15 reps):
  1a) Shoulder lift
  1b) Shoulder forward circles
  1c) Shoulder backward circles 2. Pectoral Stretch Exercise (3 sets * 10 reps; each stretch held for 30 seconds; for right and left sides) 3. Back Strengthening Exercise (3 sets * 15 reps) 4. Self Mobilization Exercise (3 sets * 10 reps; for right and left sides) 5. Cat-Camel Exercise (3 sets * 10 reps) 6. Breathing Exercises (3 sets * 10 reps): 6a) Diaphragmatic breathing 6b) Segmental breathing
  Interventions: Other: CONTROL

INTERVENTIONS:
Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — Posture exercise, stretching exercise, breathing exercise, back strengthening exercise, self-mobilization exercise, cat camel exercise and postural correction exercise will be applied.
  Arms: Intervention arm
Other: CONTROL — Posture exercise, stretching exercise, breathing exercise, back strengthening exercise, self-mobilization exercise, cat camel exercise will be applied.
  Arms: Control arm

SUMMARY:
Kyphosis-oriented exercise programs consist of isolated stretching, strengthening, and breathing exercises. However, the literature emphasizes that the body is a kinetic chain in many musculoskeletal disorders and supports holistic exercise approaches. To our knowledge, the effects of a complex exercise such as the Wall Angels exercise have not been studied in the kyphotic population. The aim of our study is to investigate whether the Wall Angels exercise combined with standard kyphosis exercises performed at home has additional effects and to contribute to the optimization of kyphosis rehabilitation programs.

DETAILED DESCRIPTION:
The study was planned as a randomized controlled double-blind study and will consist of two groups: intervention (Wall angels exercise combined with kyphosis and breathing exercises) and control (Only kyphosis and breathing exercises). The G-Power version-3.1.9 power analysis measurement method was used to determine the sample size. According to the Power Analysis conducted by taking into account the results of the studies of Elpeze and Usgu (15), it was calculated that at least 38 volunteers would be included in the study for a p<0.05 with an effect size of 0.5 and a power of 85%. The outcome measures of the study will be demographic characteristics, pain (Visual Analog Scale), trunk flexibility assessment, thoracic range of motion assessment, kyphosis index, scapula protraction, upper extremity function, respiratory capacity, postural habit and postural awareness level, and quality of life assessment. Statistical analyses will be performed using SPSS version 23.0 (IBM SPSS Statistics; IBM Corporation, Armonk, NY, USA) software. Descriptive statistics of the data will be given using mean and standard deviation for numerical variables; and percentages for qualitative variables. The Kolmogorov-Smirnov test will be used to examine the conformity of the data to normal distribution as a result of descriptive analyses. Intra-group comparisons will be evaluated using the Dependent Groups T test for groups with normal distribution, and the Wilcoxon signed ranks test for those not with normal distribution. In order to compare pre-post training values between groups, the Independent Groups T test for data with normal distribution, and the Mann Whitney-U test for data not with normal distribution will be used. The level of statistical significance will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteering to participate in the study and giving written consent
2. Being a woman/man between the ages of 18-25
3. Having a kyphotic posture

Exclusion Criteria:

1. Having a musculoskeletal disorder (scoliosis, etc.)
2. Having a neurological system disorder
3. Having a cardiopulmonary system disorder
4. Having a fracture or surgery related to the spine, rib cage, or upper extremity within the last year
5. Participating in an exercise program for kyphosis within the last 6 months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Postural Habits and Awareness Scale | From enrollment to the end of treatment at 6 weeks
  Postural habits and awareness levels will be assessed with the Postural Habits and Awareness Scale (PHAS). PHAS is a valid and reliable tool developed to assess postural habits and awareness in healthy adults. This scale consists of four sub-dimensions: postural habits and awareness, awareness of factors that impair posture, ergonomic awareness and positional awareness. PHAS is structured as a 5-point Likert scale consisting of 19 items, 7 of which are related to postural habits and 12 to postural awareness. Participants rate each item on a scale ranging from 1 (strongly disagree) to 5 (strongly agree). The total score on the scale ranges from 0 to 95, with higher scores indicating better postural habits and awareness.
Visual Analog Scale (VAS) | From enrollment to the end of treatment at 6 weeks
  The level of pain will be assessed by the participant using the Visual Analog Scale (VAS) (0: no pain; 100: unbearable pain).
Trunk Hyperextension and Lateral Flexion Flexibility Measurement | From enrollment to the end of treatment at 6 weeks
  Trunk flexibility will be measured using trunk hyperextension and lateral flexion (for right and left sides) tests and a tape measure. For the trunk hyperextension measurement, the participant is asked to stand facing the wall and with their pelvis touching the wall. First, the distance between the sternum notch and the wall is measured and recorded in this position. Then, the participant's pelvis is supported and they are asked to move their trunk backwards away from the wall. At the last point, the sternum notch and wall distance is measured again. The difference between the first and last measurements is recorded in centimeters. For the trunk lateral flexion measurement, the participant stands with their back to the wall. The tape measure is placed distal to the 3rd phalanx. The measure is recorded in centimeters. The measurement is repeated for the other side.
Flexruler Measurement (kyphosis index) | From enrollment to the end of treatment at 6 weeks
  The kyphosis index will be calculated using the appropriate formula after the measurement with the flexible ruler. The flexible ruler is a metal covered with plastic, approximately 60 cm long, which can be molded according to the contour of the spine to measure the curves in the sagittal plane. To determine the kyphosis index, the spinous processes of the C7 and T12 vertebrae are determined as references and the participant's kyphosis shape is evaluated with the flexible ruler and transferred to paper. The kyphosis index is calculated by evaluating the angle formed between the distance between C7 and T12, defined as thoracic length, and the distance of the kyphosis peak, defined as thoracic width, to the thoracic length line.
Inclinometer Tests | From enrollment to the end of treatment at 6 weeks
  Thoracic range of motion will be measured using an inclinometer for flexion and rotation (for the right and left sides). The spinous processes of the T1 and T12 vertebrae are marked as reference points. For the measurement of thoracic flexion, the inclinometer is placed vertically on the T1 vertebra and the participant is asked to lean forward so that the lumbar region does not participate in the movement. The value obtained at this point is recorded in degrees for the T1 vertebra flexion. Immediately afterwards, the inclinometer is placed vertically on the T12 vertebra and the T12 vertebra flexion is recorded in degrees. For thoracic right and left rotations, the inclinometer is placed horizontally on the T1 vertebra. The participant is asked to rotate the thoracic region and the value at the last point is recorded in degrees for the T1 vertebra. Immediately afterwards, the degree for the T12 vertebra is recorded.
Scapula Protraction Test | From enrollment to the end of treatment at 6 weeks
  For the right and left scapula, the inferior edge of the scapula is determined and the vertical distance to the midline of the spine is measured with a tape measure and recorded in centimeters.
Chest Circumference Measurement | From enrollment to the end of treatment at 6 weeks
  Respiratory capacity will be recorded in centimeters by taking the difference between the chest circumference measurements obtained at maximum inspiration and maximum expiration from the axillary, epigastric and subcostal regions. The greater the difference, the better the pulmonary function.
the Quick Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire | From enrollment to the end of treatment at 6 weeks
  The DASH is a questionnaire designed to assess disability resulting from upper extremity injuries, activity limitations, leisure activities, and work participation restrictions. The questionnaire consists of three sections. The first section contains 30 items: 21 items assessing difficulties in activities of daily living, 5 items assessing symptoms, and 4 items assessing social function, work, sleep, and self-esteem. This first section determines the Function/Symptom Model (DASH-FS) score. All questions are scored on a 5-point Likert-type scale (1: no difficulty, 5: cannot do at all) (0: no disability, 100: maximum disability). Scores range from 0 to 100 for each section (0: no disability, 100: maximum disability).
SRS22 Patient Outcome Questionnaires | From enrollment to the end of treatment at 6 weeks
  Quality of life will be assessed with the Scoliosis Research Society Patient Questionnaire. The SRS-22 is a valid and reliable scoliosis-specific quality of life scale developed by Haher et al. and modified by the Scoliosis Research Society to assess the current perception of medical status and self-image in patients with idiopathic scoliosis. The scale consists of five subscales consisting of 22 questions, including pain, general body image, spine function, mental health, and treatment satisfaction. Participants rate each question on a scale of 1 (most negative) to 5 (most positive). Scores for each subscale range from 0 to 25, while the total score for treatment satisfaction ranges from 0 to 10. Higher scores on the scale indicate improved quality of life, while lower scores reflect decreased quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mesut Ergan, asst. prof., Study Director — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University Faculty of Health Science, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No